CLINICAL TRIAL: NCT05591833
Title: Single Anastomosis Sleeve Ileal Bypass Versus Single Anastomosis Sleeve Jejunal as a Treatment of Morbid Obesity
Brief Title: Single Anastomosis Sleeve Ileal Bypass Versus Single Anastomosis Sleeve Jejunal Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, Assistant Professor & Consultant of General Surgery and laparo-endoscopy, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: fac.med 22.26
Record Dates: First submitted 2022-05-07; First posted 2022-10-24 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SASI (Active Comparator)
  Interventions: Procedure: SASI
- SAS-J (Experimental)
  Interventions: Procedure: SAS-J

INTERVENTIONS:
Procedure: SASI — Single-Anastomosis Sleeve ileal (SASI) Bypass
  Arms: SASI
Procedure: SAS-J — Single-Anastomosis Sleeve Jejunal (SAS-J) Bypass
  Arms: SAS-J

SUMMARY:
to compare the results of SASI to SAS-J in treatment of morbid obesity

DETAILED DESCRIPTION:
200 of patients indicated for obesity surgery will be divided into 2 groups : Group 1, will be operated by SASI and Group 2, will be operated by SAS-J

ELIGIBILITY:
Inclusion Criteria:

* obese patients with BMI more than 40 with or without co-morbidity or more than 35 with co-morbidity
* patients fit for laparoscopic surgery
* give approval to share in the study

Exclusion Criteria:

* patients refused to share in the study
* patients unfit for surgery
* patients aged less than 18 and older than 60
* patient with previous upper abdominal surgery either for obesity or other diseases
* revisional bariatric procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
nutritional deficiency | 12 months
  the effect of the 2 procedures on nutritional status by doing the following investigations to collectively give idea about deficiency this investigation including: Hb% ( in mg/dL), vitamin D (in ng/mL) , vitamin B ( in pg/mL), Serum Ca (in mg/dL) serum Zinc (in μg/dL) serum Iron ( in mcg/dL) serum Folate (in μg/L) and serum albumin ( in g/dL)

SECONDARY OUTCOMES:
comorbidities | 1 year
  change in comorbidities including diabetes by change in hemoglobin C level, hypertension by measuring arterial blood pressure using sphygmomanometer
complications | 1 year
  early and late complications
weight loss | 12 months
  the effect of the 2 procedures on weight measured by percentage of excess weight loss

CONTACTS AND LOCATIONS:
Locations (1):
- Minia university hospital, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided